CLINICAL TRIAL: NCT06745037
Title: Predictive Value of Blood-based Biomarkers on the Functional Outcome in Young Adult Patients with Spontaneous Intracerebral Hemorrhage
Brief Title: Interventional Study for Detection of Prognosis of Blood Based Biomarkers in Intracerebral Hemorrhage
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasmin Sherif Mosabah, Resident doctor, Assiut University
Other Study IDs: Intracerebral hemorrhage
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Intracerebral Hemorrhage
Keywords: Hemorrhage; Biomarkers; Detection
MeSH Terms: conditions — Cerebral Hemorrhage; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Young adults with intracerebral haemorrhage: Cohort prospective study for detection of blood based biomarkers of intracerebral hemorrhage in young adults.

SUMMARY:
Explore blood based biomarkers in patients with intracerebral haemorrhage [cbc. Pt. LDH.CRP. Cholesterol. Na. K.. Mg. Urea Ca. Uric acid]

DETAILED DESCRIPTION:
Spontaneous intracerebral hemorrhage (ICH) is a common subtype of stroke and accounts for nearly 10% to 30% of all strokes [1]. ICH posed a significant health burden in China in 2019, contributing to 25 million disability-adjusted life years (DALYs). It is associated with an early mortality rate of approximately 30-40% and has shown no reduction in prevalence in recent decades [2]. The higher incidence and mortality of ICH in middle-income and low-income countries may be attributed to limited public awareness regarding preventive measures, as well as challenges in accessing healthcare services [3]. So far, few treatment possibilities have yielded conclusive benefits. However, numerous predictors of poor outcomes after ICH have been suggested, including hematoma volume, hematoma expansion, perihematomal edema (PHE), and the presence and quantity of intraventricular hemorrhage growth [4,5,6,7]. Similarly, researchers continue to search for various blood-based biomarkers to guide management and predict outcomes after acute ICH [8,9,10,11,12]. A growing number of studies have shown that many novel biomarkers, such as C-reactive protein (CRP), S100A12, and interleukin-6, are associated with adverse outcomes in patients with ICH [8,9,10]. Thus, the application of blood-based biomarkers may improve risk stratification and aid clinical decisions in patients with ICH.

Therefore, in this review, we assessed the data available in the literature regarding the diagnostic and prognostic value of circulating blood biomarkers in patients with ICH. For each biomarker, we depicted the detailed characteristics in order to shed light on potential future clinical applications Intracerebral hemorrhage (ICH) is the second most common subtype of stroke and a critical disease usually leading to severe disability or death. ICH is more common in advanced age, male sex, and low- and middle-income countries. The case fatality rate of ICH is high, and only 12% to 39% of survivors can achieve long-term functional independence. Risk factors of ICH are hypertension, current smoking, excessive alcohol consumption, hypocholesterolemia, and drugs. Clinical presentation varies according to the size and location of hematoma, and intraventricular extension of hemorrhage.

ELIGIBILITY:
* Inclusion criteria:

  1. both sex
  2. Age between 25 to 40 years old.
  3. symptoms suggestive of intracerebral hemorrhage

     Exclusion criteria:

  <!-- -->

  1. Age group below 25 years and above 40 years
  2. traumatic cerebral haemorrhage
  3. extradural,subdural,subarachnoid hemorrhage
  4. Hemorrhagic infarction

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young adults patients
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
: Predictive value of blood-based biomarkers on the functional outcome in young adult patients with spontaneous intracerebral hemorrhage. | 2 years
  Explore blood based biomarkers in patients with intracerebral haemorrhage [cbc. Pt. LDH.CRP. Cholesterol. Na. K.. Mg. Urea Ca. Uric acid]
: Predictive value of blood-based biomarkers on the functional outcome in young adult patients with spontaneous intracerebral hemorrhage. | 2 years

SECONDARY OUTCOMES:
: Predictive value of blood-based biomarkers on the functional outcome in young adult patients with spontaneous intracerebral hemorrhage. | 2 years